CLINICAL TRIAL: NCT01778140
Title: Randomized Controlled Trial: Comparing Effects of Patient-Specific Versus Non-Patient-Specific Computerized Reminder System to Reduce Contrast-Induced Nephropathy
Brief Title: Comparing Effects of Patient-specific Versus Non-patient-specific Computerized Reminder System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NSC100-2320-B-038-034
Record Dates: First submitted 2012-12-26; First posted 2013-01-29 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Radiographic Contrast Agent Nephropathy
Keywords: Clinical Decision Support Systems; Contrast-induced nephropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Patient-specific reminder (Experimental): Intervention: Patient-specific computerized reminder. The physicians assigned to this arm will use the patient-specific CDSS on CPOE. The patient-specific reminder is designed as a real-time CDSS implemented on CPOE to monitor physician's contrast-enhanced image study orders. Computerized pop-up reminders provide the patient-specific CIN risk profile and optimal decision options which are generated when patients with high risk or with unknown risk of CIN are encountered.
  Interventions: Other: Patient-specific computerized reminder
- Non-patient-specific reminder (Active Comparator): Intervention: Non-patient-specific Computerized reminder. The physicians assigned to this arm will use the Non-patient-specific reminders through CPOE. Non-patient-specific reminders always pops up to remind physicians to check their patient's CIN risk no matter what CIN risk is.
  Interventions: Other: Non-patient-specific computerized reminder
- Control Arm (No Intervention): The physicians assigned to this arm will not use and any computerized reminder.

INTERVENTIONS:
Other: Patient-specific computerized reminder — The intervention targets are physicians,not patients. This CDSS alerts physicians only when the patient with high risk of contrast-induced-nephropathy(CIN) is encountered. On the contrast, the CDSS will not alert when the patient without CIN risk is encountered.
  Other Names: Patient-specific CDSS
  Arms: Patient-specific reminder
Other: Non-patient-specific computerized reminder — The non-patient-specific computerized reminder always pops up to remind physicians to check their patient's CIN risk no matter what CIN risk is.
  Other Names: Non-patient-specific CDSS
  Arms: Non-patient-specific reminder

SUMMARY:
The investigators hypothesize that a Clinical Decision Support System (CDSS) designed with "Patient-Specific" reminders yields superior performance than that with "Non-patient-specific" reminders in preventing contrast-induced nephropathy.

DETAILED DESCRIPTION:
We hypothesize that a clinical decision support system (CDSS) designed with "Patient-specific" reminders yields superior performance than that with "Non-patient-specific" reminders in preventing contrast-induced nephropathy.

A 3-arm randomized controlled trial (RCT) will be performed by cluster randomization using physicians as the unit of allocation. Physicians in 3 university medical centers will be randomly assigned into 1) patient-specific arm with Anti Contrast-Induced-Nephropathy(Anti-CIN) reminder, 2) non-patient-specific reminder arm, and 3) the control arm without any reminders, respectively.

The patient-specific alert, Anti-CIN system, is designed as a real-time CDSS implementation on CPOE for monitoring physician's contrast-enhanced CT and IVP orders. Computerized pop-up reminders provide the patient-specific encounters with optimal decision options when patients are at a high CIN risk or patients with unknown risk factors are encountered. Non-patient-specific reminders always pop up no matter whether the patient is at a high risk or not.

ELIGIBILITY:
Inclusion Criteria:

* Our intervention targets are physicians but not patients. All physicians working in the hospital may join this trial.

Exclusion Criteria:

* The physician who never orders a CT scan or IVU study will be excluded
* The physician who never operates the CPOE by himself or herself will be excluded

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
The percentage of contrast-enhanced imaging(CEI) orders with high CIN risk | Physicains who participated in this trial will be followed for an expected average of 12 months
  The number of CEI ordered for patients at high CIN risk, divided by the total number of CEI orders. [CEI]: contrast-enhanced image studies,such as CT or IVU. [CIN]: contrast-induced nephropathy

SECONDARY OUTCOMES:
The order elimination rate of high CIN risk orders attributed to the computerized reminder | Physicains who participated in this trial will be followed for an expected average of 12 months
  The number of CEI orders with high CIN risk cancelled by the physician attributed to our computerized reminder, divided by the total number of CEI orders with high CIN risk.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chuan Li, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei medical university hospital, Taipei, Taiwan